CLINICAL TRIAL: NCT02382302
Title: A Smart Phone-based Tele-consultation System in the Management of Chronic Pressure Ulcer
Brief Title: Research to Evaluate Efficiency in U-health Solution Service for the Chronic Wound Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chan-Yeong Heo (Other)
Collaborators: KT Corporation (Industry)
Responsible Party: Sponsor-Investigator, Chan-Yeong Heo, Assistant Professor, Seoul National University Hospital
Organization: Seoul National University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: E-1106/063-005
Record Dates: First submitted 2015-02-17; First posted 2015-03-06 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Pressure Ulcer
Keywords: U-health; chronic wound management
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Telemedicine system (Experimental): Telemedicine system
  Interventions: Device: Telemedicine system

INTERVENTIONS:
Device: Telemedicine system — The data such as photographs can be collected simply using built-in cameras installed in smart-phones that used the standard touch-screen user interface (UI) and camera installed in the iPhone3GS and iPhone4 using iOS 3.0 and iOS 5.0, respectively. Subjects were instructed to transmit the photographs of the wounds then investigator performed the photography in such a manner that the size of pressure ulcer should be automatically measured based on a 1 cm x 1 cm-sized indicator on the screen.

SUMMARY:
This trial is a prospective research to evaluate efficiency in U-health solution service based on Mobile for the chronic wound management.

DETAILED DESCRIPTION:
This trial conducted to assess the efficiency of teleconsultation using the smart-phone-based store-and-forward system in promoting the wound healing process as well as cost-effectiveness in patients with pressure ulcer.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have pressure ulcer
* Subjects who voluntarily decided the participation of the study and signed the informed consent

Exclusion Criteria:

* Subjects who have Osteomyelitis
* Subjects who have suppuration
* Subjects who participated in other clinical trial within 30 days from screening date

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-07; Primary Completion 2012-01 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Concordance rate for the wound and the type of dressing on the Pressure Sore Status Tool (PSST) | 4weeks post-treatment
  1. Data collection
     * The measurement of the size of pressure ulcer
     * Medical examination;the degree of recovery of pressure ulcer
  2. Remote physician monitoring
     - The patient data was transmitted from the smart-phone to the website via open application programming interface (API)
  3. Prescription
  4. Data analysis - One plastic surgeon, one Wound Ostomy Continence Nurse(WOCN) and one researcher grossly examined the wound sites of each patient and assessed the pressure ulcer using the revised PSST based on a 4-6 point scale.

SECONDARY OUTCOMES:
Concordance rate for the wound and the type of dressing on the Pressure Sore Status Tool (PSST) | 1week post-treatment
  1. Data collection
     * The measurement of the size of pressure ulcer
     * Medical examination;the degree of recovery of pressure ulcer
  2. Remote physician monitoring
     - The patient data was transmitted from the smart-phone to the website via open application programming interface (API)
  3. Prescription
  4. Data analysis - One plastic surgeon, one Wound Ostomy Continence Nurse(WOCN) and one researcher grossly examined the wound sites of each patient and assessed the pressure ulcer using the revised PSST based on a 4-6 point scale.
Concordance rate for the wound and the type of dressing on the Pressure Sore Status Tool (PSST) | 2weeks post-treatment
  1. Data collection
     * The measurement of the size of pressure ulcer
     * Medical examination;the degree of recovery of pressure ulcer
  2. Remote physician monitoring
     - The patient data was transmitted from the smart-phone to the website via open application programming interface (API)
  3. Prescription
  4. Data analysis - One plastic surgeon, one Wound Ostomy Continence Nurse(WOCN) and one researcher grossly examined the wound sites of each patient and assessed the pressure ulcer using the revised PSST based on a 4-6 point scale.
Concordance rate for the wound and the type of dressing on the Pressure Sore Status Tool (PSST) | 3weeks post-treatment
  1. Data collection
     * The measurement of the size of pressure ulcer
     * Medical examination;the degree of recovery of pressure ulcer
  2. Remote physician monitoring
     - The patient data was transmitted from the smart-phone to the website via open application programming interface (API)
  3. Prescription
  4. Data analysis - One plastic surgeon, one Wound Ostomy Continence Nurse(WOCN) and one researcher grossly examined the wound sites of each patient and assessed the pressure ulcer using the revised PSST based on a 4-6 point scale.

CONTACTS AND LOCATIONS:
Overall Officials: ChanYeong Heo, Ph.D, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea